CLINICAL TRIAL: NCT06975657
Title: Community-engaged Research to Promote Mental Health and Successful Reentry Outcomes Following Incarceration
Brief Title: Well-being Skills for Reentry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1269; A483000 (Other: UW Madison); Protocol Version 12/10/2025 (Other: UW Madison)
Record Dates: First submitted 2025-05-07; First posted 2025-05-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Formerly Incarcerated Adults

STUDY DESIGN:
Intervention Model Description: The groups will be randomized to one of two groups in a 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Wellbeing skills training (Experimental)
  Interventions: Behavioral: Wellbeing skills for reentry; Device: Healthy Minds Program
- Waitlist control (No Intervention)

INTERVENTIONS:
Behavioral: Wellbeing skills for reentry — An 8-week, in-person meditation training program for formerly incarcerated adults, with practices and concepts grounded in the four pillars of the Healthy Minds Program (awareness, connection, insight, and purpose) that are supported by custom meditation practices presented in the Healthy Minds Program App.
  Arms: Wellbeing skills training
Device: Healthy Minds Program — A customized version of the Healthy Minds Program app will allow participants to listen to recorded meditation practices in support of the in-person curriculum.
  Arms: Wellbeing skills training

SUMMARY:
The goal of this clinical trial is to learn if a mindfulness skills training program has mental health benefits for people returning to the community following incarceration. The main questions it aims to answer are:

* Does mindfulness skills training improve symptoms of anxiety and depression?
* Do participants find this mindfulness program to be acceptable and feasible to participate in?

Researchers will compare outcomes for participants in the mindfulness training program to those in a waitlist control group who will receive the mindfulness program after the end of the study.

Participants will:

* Complete an initial intake visit, consisting of an interview and questionnaires
* Randomly be assigned to a mindfulness group or a waitlist control group
* Participate in weekly mindfulness classes for 6 weeks (mindfulness group only)
* Complete a set of questionnaires after the conclusion of the mindfulness classes
* Complete a set of questionnaires and an interview 2 months after the conclusion of the mindfulness classes

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Formerly incarcerated in a local jail, state or federal prison
* Can read, speak and understand English
* Able to provide informed consent

Exclusion Criteria:

* Suicidal ideation with some intent to act or with a specific plan and intent
* Active psychosis
* Daily or nearly daily use (over the past 3 months) of the following substances: cocaine, amphetamines, inhalants, sedatives or sleeping pills, hallucinogens, or opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Psychological distress | Baseline, following week 8 of intervention period (approximately 10 weeks), 2-month follow-up after intervention period (approximately 18 weeks)
  Standardized composite score of three common data elements: the Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder-7 (GAD-7), and Perceived Stress Scale-4 (PSS-4). To generate a composite psychological distress measure, PHQ-9, GAD-7, and PSS-4 scores will be z-transformed and then averaged. Resulting composite distress scores will have a mean of 0 and SD of 1, with higher scores indicating greater distress.
Feasibility based on Theoretical Framework of Acceptability (TFA) questionnaire | Following week 8 of intervention period (approximately 10 weeks)
  TFA is an 8 item questionnaire, which uses a 5-point Likert scale to assess acceptability of the intervention. Scores range from 8-40, with higher scores indicating greater acceptability.

SECONDARY OUTCOMES:
Change in Awareness | Baseline, following week 8 of intervention period (approximately 10 weeks), 2-month follow-up after intervention period (approximately 18 weeks)
  Change in awareness will be measured using the Five Facet Mindfulness Questionnaire (FFMQ) Act with Awareness. The FFMQ is an 8 item questionnaire and is scored on a 5-pooint Likert scale. Scores range from 8-40, with higher scores indicating a lower sense of awareness.
Change in Connection | Baseline, following week 8 of intervention period (approximately 10 weeks), 2-month follow-up after intervention period (approximately 18 weeks)
  Change in Connection will be measured using the Perceived Isolation questionnaire, which is a 9 item questionnaire. Each of the 9 items is standardized. The standardized scores for the 9 items are then averaged to create a single Perceived Isolation score. A higher average score means the individual experiences more perceived isolation or loneliness.
Change in Insight | Baseline, following week 8 of intervention period (approximately 10 weeks), 2-month follow-up after intervention period (approximately 18 weeks)
  Change in Insight will be measured using scores of Metacognitive Process of Decentering, which is a 15 item questionnaire. It is scored on a 5-point Likert scale, with scores ranging from 15-75. Lower scores indicate lower levels of insight.
Change in Purpose | Baseline, following week 8 of intervention period (approximately 10 weeks), 2-month follow-up after intervention period (approximately 18 weeks)
  Change in purpose will be measured using the NIH Toolbox Meaning & Purpose. The Toolbox is a 4 item questionnaire and is scored on a 5-pooint Likert scale. Scores range from 4-20, with higher scores indicating a greater sense of purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Grupe, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes